CLINICAL TRIAL: NCT02040038
Title: Diabetes Self-Management & Support LIVE (Learning in Virtual Environments)
Brief Title: Diabetes Self-Management & Support LIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00043325; 1R01HL118189-01 (NIH)
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Virtual Environment; Self-Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LIVE Arm (Experimental): Participation in 3D virtual environment for DSMT/S for a period of 12 months.
  Interventions: Behavioral: LIVE
- Website (Active Comparator): Participation in 2D website for DSMT/S for a period of 12 months.
  Interventions: Behavioral: Website

INTERVENTIONS:
Behavioral: LIVE — 3-D Virtual Environment for DSMT/S
  Arms: LIVE Arm
Behavioral: Website — 2-D Website participation for DSMT/S
  Arms: Website

SUMMARY:
The purpose of this study is to determine whether participation in virtual environment which incorporates real-time diabetes self management and support (DSMT/S) is associated with positive changes in behavior and metabolic outcomes as compared to traditional web-based DSMT/S.

ELIGIBILITY:
Inclusion Criteria:

* Live in close proximity to Duke University Medical Center (DUMC) or NYU Endocrinology Clinic, or Faculty Practice and Bellevue Medical Center to facilitate follow-up research appointments
* Diagnosis of Type 2 Diabetes (T2D)
* >= 21 years old
* able to read and understand English
* access to a computer with broad band internet connection in a private location
* reachable by telephone
* no pre-existing medical condition(s) or severe diabetes related complications that would interfere with study participation (e.g.
* Are able to travel to a clinical lab for blood work

Exclusion Criteria:

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2014-07; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in Dietary Intake | 18 months
  Dietary (fat intake, fruit and vegetable intake) will be assessed at start of the study and at 3, 6, 12 and 18 months
Change in Physical Activity | 18 months
  Changes in physical activity will be measured using the Fitbit physical activity monitoring at 3, 6, 12, and 18 months.

SECONDARY OUTCOMES:
Change in HbA1C level | 18 months
  Metabolic control (HbA1c) levels will be measured at the start of the study and again at 6, 12, and 18 months
Change in BMI | 18 months
  BMI will measured at the start of study and at 6, 12, and 18 months.
Change in Waist Circumference | 18 months
  Waist circumference will be measured at start of study and at 6, 12, and 18 months.
Change in Blood Pressure | 18 months
  Blood pressure will be measured at the start of the study and again at 6, 12, and 18 months.
Change in Lipid Levels | 18 months
  High density lipoprotein (HDL), low density lipoprotein (LDL), total cholesterol (TC) and triglyceride levels will be measured at the start of the study and again at 6, 12 and 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Constance M. Johnson, PhD, Principal Investigator — Duke University School of Nursing; Allison Vorderstrasse, DNSc, Principal Investigator — Duke University School of Nursing; Gail Melkus, EdD, Principal Investigator — New York University
Locations (2):
- United States (2):
  - New York University, New York, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Johnson CM, D'Eramo Melkus G, Reagan L, Pan W, Amarasekara S, Pereira K, Hassell N, Nowlin S, Vorderstrasse A. Learning in a Virtual Environment to Improve Type 2 Diabetes Outcomes: Randomized Controlled Trial. JMIR Form Res. 2023 Apr 20;7:e40359. doi: 10.2196/40359. PMID 36962700
- [Derived] Johnson CM, McIlwain S, Gray O, Willson B, Vorderstrasse A. Creating a sustainable collaborative consumer health application for chronic disease self-management. J Biomed Inform. 2017 Jul;71:198-206. doi: 10.1016/j.jbi.2017.06.004. Epub 2017 Jun 6. PMID 28600025
- [Derived] Vorderstrasse AA, Melkus GD, Pan W, Lewinski AA, Johnson CM. Diabetes Learning in Virtual Environments: Testing the Efficacy of Self-Management Training and Support in Virtual Environments (Randomized Controlled Trial Protocol). Nurs Res. 2015 Nov-Dec;64(6):485-93. doi: 10.1097/NNR.0000000000000128. PMID 26505161